CLINICAL TRIAL: NCT05479435
Title: Comparison Effects Of Blue Prescription Program, Home Exercise Program And Supervised Exercise Approaches On Type 2 Diabetic Women
Brief Title: Comparison Effects Of Different Exercise Approaches On Type 2 DM Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, aabalay, phd student, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10840098-604.01.01-E.14291
Record Dates: First submitted 2022-01-26; First posted 2022-07-29 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized control trial with statistic analyst blind
Masking Description: We will mask only person who will do statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blue Prescription Group (Experimental): Participants will receive an exercise program designed according to their needs, desires, and abilities. They will perform the desired exercise program three days a week and will have an interview for motivation and/or modifying the program one day a week. They will also keep an activity diary.
  Interventions: Behavioral: Blue Prescription Exercise Program
- Video Based Home Exercise Group (Active Comparator): Participants will receive videos through various channels. They will perform exercises three days a week. The investigator will call them to inquire whether they are following the program or not. Additionally, they will keep an activity diary.
  Interventions: Behavioral: Video Based Home Exercise Program
- Supervised Exercise Group (Active Comparator): Participants will perform an exercise program 3 days a week under the guidance of a physiotherapist. Each group will consist of a maximum of 10 people.
  Interventions: Behavioral: Supervised Group Exercise Program

INTERVENTIONS:
Behavioral: Blue Prescription Exercise Program — After the evaluation, participants will receive feedback and physical activity training, along with an explanation of the benefits of exercise, provided in the form of a brochure. They will then be enrolled in the Blue Prescription program, which includes weekly follow-ups for 12 weeks and a re-evaluation at the end of the 12th week. Motivation and support will be offered in accordance with the Blue Prescription philosophy, addressing home exercise programs, physical activity selection, and overcoming obstacles. Participants will be encouraged to determine the most suitable program for themselves and maintain an activity diary.
  Throughout the study, participants will have the opportunity to communicate with the physiotherapist via various methods such as phone, SMS, or email.
  Arms: Blue Prescription Group
Behavioral: Video Based Home Exercise Program — After the evaluation, DM and physical activity training will be given, the benefits of exercise will be explained and these will be given as a brochure. A video exercise program will be given in the format and method desired by the participant. It will be evaluated again at the end of the 12th week.
  Arms: Video Based Home Exercise Group
Behavioral: Supervised Group Exercise Program — DM and physical activity training will be given after the assessment, the benefits of the exercise will be explained and these will be given as a brochure. Participants will engage in exercises with a physiotherapist three days a week for 12 weeks, and the effectiveness of the program will be re-evaluated at the end of the 12th week.
  Arms: Supervised Exercise Group

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) is one of the most common metabolic diseases with a complex, multifactorial etiology, and is a chronic disease with various clinical and biochemical manifestations. It has been known for a long time that T2DM treatments include medication, diet, and exercise. Exercise can improve blood glucose control, increase insulin sensitivity, respiratory capacity, well-being and cognitive functions, regulate lipid profile, blood pressure, reduce cardiovascular disease risk, abdominal obesity, weight. Although there are many studies in the literature on the effects of exercise in T2DM, there is no consensus on which exercise protocol is more effective. In the studies, the obstacles in front of the diabetic patients' adaptation to exercise; laziness, lack of motivation and energy, embarrassment from family and social environment, lack of support, time constraints, financial problems, lack of space to exercise, fear of hypoglycaemia, pain, stiffness, fatigue, shortness of breath, presence of additional diseases, fear of injury. Blue Prescription (BP) is a model developed to facilitate the participation in physical activity. In traditional home programs, patients are told what to do. The BP approach, on the other hand, involves providing the person with options for physical activity, removing the barriers to activity instead of the classical home exercise program or physical activity counselling, and being in communicate according to the person's preferences during this process. This approach has been developed to facilitate participation in physical activity and to ensure the sustainability of physical activity in individuals with chronic diseases. Philosophy of the approach aims to increase the activity level gradually, improve the quality of life and participation in the activity with motivational interview, continuous support, communication and activity diary, instead of recommending physical activity with classical methods due to the different needs, desires and preferences of people. Studies using the BP in the literature have focused on Multiple Sclerosis and stroke, and no publications on other chronic diseases have been found. The aim of this study is to examine the effects of BP, video-based home exercise and supervised group exercises on HbA1c, physical activity level, functional capacity and other metabolic control variables in primary care women with T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Between 25-65 years of age
2. Having Type 2 DM for at least 5 years
3. HbA1c value> 6.5% / Fasting blood glucose> 126 mg / dl
4. Ability to walk independently
5. Volunteering to participate in research

Exclusion Criteria:

1. Type 1 DM
2. Using insulin
3. Orthopedic and neurological diseases that prevent exercise
4. Having cardiovascular, pulmonary and systemic diseases in which exercise is contraindicated.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 1st 2021 started day. The study location was Balikesir Provincial Health Directorate, Edremit District Health Directorates Healthy Life Center, Balikesir, Turkey.
Pre-assignment Details: The participiants who diagnosed with Diabetes Mellitus Type 2, were recruited from Balikesir Provincial Health Directorate, Edremit District Health Directorates Healthy Life Center.
  They were 60 people who were assigned to the groups.
Groups:
- Blue Prescription Group: Participants will get an exercise program, which is designed by their needs, desires and abilities. They will perform a desired exercise program 3 days a week and they will make an interview for motivation and/or modifying the program one day a week. They will write an activity diary.
  Blue Prescription Exercise Program: After the evaluation, DM and physical activity training will be given, the benefits of exercise will be explained and these will be given as a brochure. It will be followed up with the blue prescription program once a week for 12 weeks and will be re-evaluated at the end of the 12th week. Motivation and support will be provided according to the blue prescription philosophy, home exercise program, physical activity selection, obstacles to the activity are discussed, the participant will be asked to determine the appropriate program and keep an activity diary. Throughout the study, the participant will be able to communicate with the physiotherapist by any method (phone, SMS, email).
- Video Based Home Exercise Group: Participants will get videos by different ways (closed link youtube, whatsapp, flash driver etc.). They will perform exercises 3 days a week. İnvestigator will phone them to ask whether they do the program or not. They will write an activity diary.
  Video Based Home Exercise Program: After the evaluation, DM and physical activity training will be given, the benefits of exercise will be explained and these will be given as a brochure. A video exercise program will be given in the format and method desired by the participant. It will be evaluated again at the end of the 12th week.
- Supervised Exercise Group: Participants will perform an exercise program 3 days a week with a physiotherapist. The group will be held maximum 10 people.
  Supervised Group Exercise Program: DM and physical activity training will be given after the assessment, the benefits of the exercise will be explained and these will be given as a brochure. Exercises will be done with a physiotherapist for 12 weeks 3 days a week and will be evaluated again at the end of the 12th week.
Period: Overall Study
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Started | 20 | 20 | 20
Completed | 19 | 20 | 18
Not Completed | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Covid 19 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.68 (9.08) | 48.85 (8.79) | 50.39 (8.46) | 50.61 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: From blue prescription group, one participant had took COVID 19, from supervised group, one participant had took COVID 19 and the other wanted to drop off by herself. So we drop off them.
  Participants
    Female | 20 | 20 | 20 | 60
    Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Hemoglobin Change
Description: Hemoglobin A1c is a blood test used to measure the effectiveness of treatment in diabetes, and sometimes to diagnose diabetes. The generally accepted reference range for Hemoglobin A1c (HbA1c) is between 4% and 6%.
Time Frame: Change from Baseline Glycosylated Hemoglobin at 12 weeks.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Groups:
- Blue Prescription Group: Participants will receive an exercise program tailored to their needs, desires, and abilities. They will engage in this program three days a week and participate in motivational interviews or program modification sessions once a week. Additionally, they will maintain an activity diary.
  As part of the Blue Prescription Exercise Program, participants will undergo an evaluation followed by diabetes and physical activity training. They will also receive a brochure explaining the benefits of exercise. The Blue Prescription program will be followed once a week for 12 weeks, with a re-evaluation at the end of this period. Motivation and support will align with the Blue Prescription philosophy, incorporating a home exercise program, discussing physical activity selection, and addressing obstacles. Participants will be encouraged to determine the most suitable program and keep an activity diary. Throughout the study, participants will have the option to communicate with the physiotherapist via phone, SMS, or email.
- Video Based Home Exercise Group: Participants will receive videos through various channels for their exercise program. They will engage in these exercises three days a week. An investigator will contact them via phone to inquire whether they are following the program. Additionally, participants will maintain an activity diary.
  Video-Based Home Exercise Program: Following an evaluation, participants will receive training on diabetes management and physical activity. They will be provided with a brochure explaining the benefits of exercise. The exercise program will be delivered in video format, tailored to the participant's preferences and chosen method of delivery. A re-evaluation will be conducted at the end of the 12th week
- Supervised Exercise Group: Participants will engage in a supervised group exercise program led by a physiotherapist, with a maximum of 10 people per group. Following an assessment, participants will receive training on diabetes management and physical activity. The benefits of exercise will be explained and provided in brochure format.
  The supervised group exercise sessions will take place three days a week for a duration of 12 weeks. At the end of the 12-week period, participants will undergo a re-evaluation.
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
percentage of glycosylated hemoglobin
  Baseline | 6.82 (1.21) | 7.17 (2.37) | 6.80 (0.94)
  At the end of 12 weeks | 6.33 (0.94) | 6.69 (2.08) | 6.32 (0.91)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.830, Kruskal-Wallis

2. Primary Outcome: Physical Activity Level Change
Description: The questionnaire provides information about the time spent by the individual in light, moderate, and vigorous activities and sitting in the last 7 days. The MET-min / week score is obtained by multiplying the MET value (metabolic equivalent) by days and minutes for each activity level. Physical activity levels are classified as:
  Physically inactive (<600 MET-min / week), Low physical activity (600-3000 MET-min / week), and Adequate physical activity (> 3000 MET-min / week). A higher score is associated with a higher physical activity level.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks)
Measure: Mean (Standard Deviation); unit: MET-min / week
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
MET-min / week
  baseline | 846.45 (615.04) | 797.20 (635.14) | 909.64 (699.90)
  at the end of the 12 weeks | 1960.89 (735.78) | 1654.05 (770.22) | 2370.11 (772.45)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.654, ANCOVA

3. Primary Outcome: Functional Capacity Change With Timed Up And Go Test
Description: The participant will sit on a chair without armrests, stand up with the command to start, walk 3 meters towards the designated point, turn around and walk to the starting point again and sit. The test is repeated 3 times and the average is taken. The time will be recorded in seconds. As time increases, the risk of falling increases.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks)
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
second
  baseline | 10.64 (1.80) | 10.31 (1.74) | 10.62 (1.71)
  at the end of the 12 weeks | 9.21 (1.29) | 8.99 (1.51) | 9.26 (1.37)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.803, ANCOVA

4. Primary Outcome: Functional Capacity Change With 6-minute Walking Test
Description: It will be performed in a 30 meter long corridor or in an open area. The participant will be asked to walk without running at the highest speed for 6 minutes. Before and during the march, the participant will be verbally encouraged and motivated. How many meters they walked will be recorded as a result of the test. Six-minute walk test results can be interpreted as follows:
  Normal: more than 500 meters Light restriction: 400 to 500 meters Moderate restriction: 300 to 400 meters Severe restriction: between 200 - 300 meters Serious restriction: less than 200 meters.
Time Frame: Change from Baseline 6-minute Walking Test Results at 12 weeks.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
meter
  baseline | 402.57 (38.52) | 405.95 (44.84) | 416.97 (49.66)
  at the end of the 12 weeks | 462.82 (44.38) | 457.85 (55.35) | 483.44 (55.32)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.398, ANCOVA

5. Primary Outcome: Fasting Plasma Glucose
Description: Measured level of glucose in the blood after 8 to 12 hours of fasting. The unit of measurement is mg/dL, the reference range is 70-110 mg/dL.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: (mg/dL)
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
(mg/dL)
  baseline | 138.21 (34.49) | 157.05 (60.90) | 128.33 (25.02)
  at the end of the 12 weeks | 115.53 (22.48) | 145.50 (43.73) | 118.28 (20.57)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.132, Kruskal-Wallis

6. Primary Outcome: High Density Lipoprotein
Description: It takes part in the transport of cholesterol from tissues and vessels to the liver and in the synthesis of vitamin D. The unit of measurement is mg/dL, the reference range is 30-96 mg/dL.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
mg/dL
  baseline | 52.74 (11.11) | 54.30 (10.31) | 54.83 (20.80)
  at the end of the 12 weeks | 59.05 (11.26) | 59.20 (10.50) | 62.53 (19.23)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.991, Kruskal-Wallis

7. Primary Outcome: Low Density Lipoprotein
Description: It provides the transport of cholesterol synthesized in the liver to the tissues and blood vessels. The unit of measurement is mg/dL, the reference range is 0- 130 mg/dL.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
mg/dL
  baseline | 136.58 (33.62) | 123.45 (24.57) | 156.00 (67.90)
  at the end of the 12 weeks | 125.37 (31.55) | 116.90 (20.79) | 130.33 (39.47)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.278, Kruskal-Wallis

8. Primary Outcome: Total Cholesterol
Description: Total cholesterol is a value that shows the total amount of cholesterol in the blood. In addition to LDL and HDL, triglyceride levels are also used to calculate total cholesterol. The unit of measurement is mg/dL, the reference range is 70-200 mg/dL.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
mg/dL
  baseline | 219.21 (46.28) | 208.40 (33.36) | 221.28 (31.84)
  at the end of the 12 weeks | 203.00 (43.61) | 189.90 (28.55) | 200.61 (27.89)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.479, ANCOVA

9. Primary Outcome: Triglyceride
Description: It is a storage nutrient molecule formed by the combination of fatty acids and glycerol molecules, which form the structure of fats in foods. The unit of measurement is mg/dL, the reference range is 0-250 mg/dL.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
mg/dL
  baseline | 173.16 (58.50) | 172.15 (36.08) | 203.12 (139.64)
  at the end of the 12 weeks | 156.00 (54.29) | 152.85 (38.48) | 184.22 (109.60)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.849, Kruskal-Wallis

10. Primary Outcome: C-reactive Protein
Description: It is a protein produced in the liver. It is a protein that is produced by cells and secreted into the blood when the body reacts to conditions such as infection, tumor, trauma, and undertakes various biochemical tasks. The unit of measurement is mg/dL, the reference range is 0-0.5 mg/dL.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
mg/dL
  baseline | 2.31 (3.63) | 1.55 (1.25) | 3.51 (4.12)
  at the end of the 12 weeks | 1.83 (2.95) | 1.51 (1.03) | 2.46 (2.55)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.504, Kruskal-Wallis

11. Primary Outcome: Systolic Blood Pressure
Description: Blood pressure is the pressure that builds up in the blood vessels when the heart contracts. It is measured with a sphygmomanometer. The cuff is placed 2.5 to 3 cm above the inside of the elbow. The stethoscope is placed under the cuff and pressed lightly. The sphygmomanometer cuff is then inflated to 20 to 30 mmHg above the level at which the pulse disappears. The control valve should be opened slightly, and air should be vented at a rate of 2-4 mmHg per second. The first sound heard as the air is released determines the systolic blood pressure. The reference range averages 120 - 130 mmHg.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
mmHg
  baseline | 128.63 (8.32) | 129.05 (8.25) | 134.78 (7.80)
  at the end of the 12 weeks | 123.63 (7.82) | 126.30 (7.76) | 129.17 (6.40)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.017, ANCOVA

12. Primary Outcome: Diastolic Blood Pressure
Description: The pressure that builds up in the blood vessels as the heart relaxes is known as diastolic blood pressure. It is measured using a sphygmomanometer, which is placed 2.5 to 3 cm above the inside of the elbow. The stethoscope is placed under the cuff and lightly pressed. The sphygmomanometer cuff is then inflated to 20 to 30 mmHg above the point where the pulse disappears. The control valve should be opened slightly, and air should be released at a rate of 2-4 mmHg per second. The point at which the sound becomes inaudible is considered the diastolic blood pressure. The reference range averages 70 - 90 mmHg.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
mmHg
  baseline | 77.05 (8.08) | 80.10 (6.16) | 83.50 (6.72)
  at the end of the 12 weeks | 75.47 (7.24) | 78.85 (6.01) | 81.39 (6.43)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.025, Kruskal-Wallis

13. Primary Outcome: Heart Rate
Description: It is the value that shows how many times the heart beats in a minute. Measurement from the wrist: measured from the radial artery with 3 fingers with the palm facing up. The reference range is between 60 and 100 beats per minute (bpm).
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
beats/min
  baseline | 72.63 (7.30) | 73.70 (6.28) | 76.56 (5.55)
  at the end of the 12 weeks | 71.16 (6.10) | 72.30 (5.11) | 74.11 (4.20)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.016, ANCOVA

14. Secondary Outcome: Body Fat Ratio Change With Bioelectrical Impedance Analysis (BIA)
Description: -Bioelectrical Impedance Analysis (BIA): The basic principle is to measure the impedance by using the resistance and conductivity that a very small amount of electrical current encounters when passing through tissues. Reference values for Bioelectrical Impedance Analysis (BIA) may vary depending on factors such as age, gender, height and weight. However, a typical BIA reference range for generally healthy adults is as follows:
  Body Fat Percentage:
  For women: 20% - 25%
  Body Mass Index (BMI):
  Normal Range: 18.5 - 24.9 kg/m² However, these values can vary greatly between individuals and may vary depending on many factors such as clinical conditions, lifestyle factors, ethnicity, etc. Therefore, BIA results should be interpreted taking into account the individual's personal health status and goals. "Tanita SC-330" brand device will be used in our study.
Time Frame: Change from Baseline Bioelectrical Impedance Analysis at 12 weeks.
Measure: Mean (Standard Deviation); unit: percent body fat
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
percent body fat
  baseline | 43.63 (4.86) | 40.27 (4.53) | 43.54 (4.04)
  at the end of the 12 weeks | 41.79 (5.04) | 38.30 (4.77) | 41.06 (4.15)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.041, ANCOVA

15. Secondary Outcome: Body Fat Ratio Change With Skinfold Analysis
Description: All measurements will be made on the right side of the body. The caliper will be placed approximately 1 cm from the thumb and index finger, and 1-2 seconds will be waited before the caliper is read. Body fat percentages of individuals will be calculated using Jackson-Pollock 7 region equations; Triceps, Subscapularis, Midaxillary, Abdominal, Chest, Suprailiac. The Jackson-Pollock skinfold thickness method is a method used to estimate body fat percentage. Reference values may vary depending on factors such as the person's gender, age range and lifestyle. However, in general, reference values for body fat percentage obtained using the Jackson-Pollock formula are as follows:
  Athletic women: 14-20% Women in good shape: 21-24% Average women: 25-31% Overweight women: 32-39% Obese women: 40% and above
Time Frame: Change from Baseline Skinfold Analysis at 12 weeks.
Measure: Mean (Standard Deviation); unit: percent body fat
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
percent body fat
  baseline | 42.76 (3.04) | 41.59 (3.39) | 43.36 (1.95)
  at the end of the 12 weeks | 41.85 (3.19) | 40.78 (3.36) | 42.55 (2.10)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.352, Kruskal-Wallis

16. Secondary Outcome: Flexibility Change With Fingertip-to-floor Distance Measure
Description: During the test, the participant will be asked to lean forward without bending their knees and try to touch the fingertip. The distance between the tip of the third finger of the hand and the ground will be measured and the result will be recorded in cm. This distance is considered normal up to 0 cm in women and up to 10 cm in men.
Time Frame: Change from Baseline Fingertip-to-floor Distance Measure at 12 weeks.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
centimeter
  baseline | 9.05 (4.08) | 10.90 (8.90) | 9.67 (5.79)
  at the end of the 12 weeks | 4.16 (4.51) | 7.70 (7.23) | 5.67 (4.28)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.390, Kruskal-Wallis

17. Secondary Outcome: Flexibility Change With Trunk Lateral Flexion Measure
Description: The participant will be asked to stand with their feet slightly open, parallel to each other, arms next to the trunk. Mark the distal end of the third finger of the hand on the thigh, and the participant will be asked to perform lateral flexion. The point where the distal of the third finger comes from is marked again. The distance between the two points is cm. will be recorded in terms. A higher value is associated with good flexibility.
Time Frame: Change from Baseline Trunk Lateral Flexion Measure at 12 weeks.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
centimeter
  baseline | 12.95 (3.31) | 13.68 (4.19) | 12.61 (3.50)
  at the end of the 12 weeks | 17.47 (3.29) | 17.15 (4.22) | 18.89 (2.91)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.928, ANCOVA

18. Secondary Outcome: Life Quality
Description: The Diabetes Quality of Life (DQoL) Questionnaire consists of 46 items divided into four subscales: Satisfaction (15 items), Impact (20 items), Worry - Social/Vocational (7 items), and Worry - Diabetes-Related (4 items). Each item is rated on a 5-point Likert scale ranging from 1 to 5. Depending on the item, higher scores may indicate either greater dissatisfaction, greater impact, or higher worry. Subscale scores are calculated by summing item responses within each subscale. The total score is the sum of all items and ranges from 46 to 230. Higher total scores indicate a lower diabetes-related quality of life.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
units on a scale
  baseline | 3.57 (0.58) | 3.61 (0.51) | 3.61 (0.45)
  at the end of the 12 weeks | 4.31 (0.33) | 4.29 (0.30) | 4.60 (0.24)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.558, Kruskal-Wallis

19. Secondary Outcome: Depression
Description: It will be evaluated with the Beck Depression Scale. The scale is used to measure the level of depression with a 21-item multiple-choice question. Each question is evaluated within a certain score range, and the total score shows the person's depression level. However, the scale does not have an official "reference" range because scoring may vary depending on clinical or research purposes.
  In general, Beck Depression Inventory (BDI) scores can be interpreted as follows:
  0-13 points: Mild or minimal depression 14-19 points: Mild depression 20-28 points: Moderate depression 29-63 points: Severe depression
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
units on a scale
  baseline | 12.95 (7.42) | 13.15 (4.66) | 16.17 (5.22)
  at the end of the 12weeks | 9.37 (5.24) | 9.65 (4.13) | 9.78 (4.41)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.133, Kruskal-Wallis

20. Secondary Outcome: Contentment
Description: It will be evaluated with The Diabetes Treatment Satisfaction Questionnaire (DTSQ). The questionnaire measures how the individual perceives glycemic control and satisfaction with the treatment. Suitable for Type 1 DM and Type 2 DM. It consists of 8 items and is scored on a 0-6 Likert scale. 6 items 1, 4, 5, 6, 7, 8); It meets to determine satisfaction between 0 (not at all) and 6 (very satisfied). Of the remaining items, 2, 0 (never) to 6 almost always) measure the frequency of detection of hyperglycemia, and item 3 measures the frequency of detecting hypoglycemia. The highest score is calculated as 36. High scores indicate satisfaction with treatment, while low scores indicate dissatisfaction.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
units on a scale
  baseline | 21.37 (4.03) | 22.30 (4.73) | 19.28 (4.90)
  at the end of the 12 weeks | 29.63 (2.03) | 29.75 (2.65) | 32.17 (1.58)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.367, Kruskal-Wallis

21. Secondary Outcome: Height
Description: It will be measured with a stadiometer. Head, shoulders, back, hips, calves and heels will touch the stadiometer, stand upright with feet shoulder-width apart, slide of height meter will be pulled down.
Time Frame: In the beginning of the intervention
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
meter | 1.57 (0.06) | 1.58 (0.05) | 1.59 (0.05)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.631, ANCOVA

22. Secondary Outcome: Weight
Description: It will be measured with a standard weighing instrument.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
kg
  baseline | 88.55 (12.81) | 79.87 (11.65) | 87.93 (13.14)
  at the end of the 12 weeks | 84.69 (10.86) | 77.96 (11.07) | 81.40 (11.82)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.056, ANCOVA

23. Secondary Outcome: Neck Circumference
Description: In the anatomical position, the tape measure is measured just below the thyroid cartilage.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
centimeter
  baseline | 38.13 (2.80) | 38.05 (3.02) | 38.53 (2.84)
  at the end of the 12 weeks | 37.05 (2.46) | 36.95 (2.82) | 36.83 (2.15)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.979, ANCOVA

24. Secondary Outcome: Waist Circumference
Description: It is measured at the thinnest point between the lowest rib and anterior superior to the processus spina ilica in the anatomical position.
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
centimeter
  baseline | 104.42 (14.45) | 103.10 (12.54) | 109.56 (10.26)
  at the end of the 12 weeks | 100.16 (13.00) | 98.60 (12.65) | 102.78 (8.02)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.377, ANCOVA

25. Secondary Outcome: Hip Circumference
Description: Measured at the widest point of the Gluteus Maximus muscle in the anatomical position
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
centimeter
  baseline | 120.58 (12.13) | 113.60 (7.96) | 116.72 (8.72)
  at the end of the 12 weeks | 117.84 (11.33) | 111.90 (7.97) | 112.17 (7.83)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.979, ANCOVA

26. Secondary Outcome: Body Mass Index (BMI)
Description: BMI will be calculated by dividing body weight (kg) by height square (m^2). General reference ranges for BMI are as follows:
  If BMI is less than 18.5 kg/m^2: Underweight If BMI is between 18.5-24.9 kg/m^2: Normal weight If BMI is between 25.0-29.9 kg/m^2: Overweight If BMI is 30.0 kg/m^2 and above: Obese
Time Frame: In the beginning of the intervention and at the end of the exercise program (12 weeks).
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
Number analyzed (Participants) | 19 | 20 | 18
kg/m^2
  baseline | 35.93 (5.73) | 32.04 (5.04) | 34.76 (5.03)
  at the end of the 12 weeks | 34.36 (4.95) | 31.24 (4.74) | 32.32 (4.53)
Statistical Analysis 1: Comparison: Blue Prescription Group vs Video Based Home Exercise Group vs Supervised Exercise Group; Test type: Other; p = 0.055, ANCOVA

ADVERSE EVENTS:
Time Frame: 2 years
Description: They were no any adverse event.
Arm/Group | Blue Prescription Group | Video Based Home Exercise Group | Supervised Exercise Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT05479435/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT05479435/SAP_001.pdf
  • Informed Consent Form (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT05479435/ICF_002.pdf